CLINICAL TRIAL: NCT01260883
Title: Ketorolac in Postoperative Infants: Pharmacokinetics and Safety
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Anne M. Lynn, Professor, Anesthesiology and Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IND 59883; NCT00014716 (obsolete NCT alias)
Record Dates: First submitted 2010-12-09; First posted 2010-12-15 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Postoperative Pain in Infants
Keywords: ketorolac pharmacokinetics; ketorolac stereo-isomers; infants; postoperative analgesia; safety
MeSH Terms: interventions — Ketorolac Tromethamine; Glucose; Water

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ketorolac 1 mg/kg (Experimental): ketorolac 1 mg/kg iv given by 10 min infusion
  Interventions: Drug: Ketorolac Tromethamine 1 mg/kg
- ketorolac 0.5 mg/kg (Active Comparator): ketorolac 0.5 mg/kg iv given by 10 min infusion
  Interventions: Drug: Ketorolac Tromethamine 0.5 mg/kg
- placebo (Sham Comparator): placebo group received D5W 10 min infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine 1 mg/kg — Ketorolac Tromethamine 1 mg/kg infusion over 10 minutes intravenous (IV) infusion. Blood sampling in for up to 12 hours after infusion for analysis of ketorolac concentrations and safety assessments.
  Other Names: toradol
  Arms: ketorolac 1 mg/kg
Drug: Ketorolac Tromethamine 0.5 mg/kg — Ketorolac Tromethamine 0.5 mg/kg infusion over 10 minutes intravenous (IV) infusion. Blood sampling for up to 12 hours after infusion for analysis of ketorolac concentrations and safety assessments.
  Other Names: toradol
  Arms: ketorolac 0.5 mg/kg
Drug: Placebo — Dextrose in water (D5W) infusion over 10 minutes intravenous (IV) infusion. Blood sampling for up to 12 hours after infusion for analysis of ketorolac concentrations and safety assessments.
  Other Names: Dextrose in water (D5W)
  Arms: placebo

SUMMARY:
Infants handle ketorolac differently than adults. Study of handling of this pain medication given to infants following surgery. Detailed analysis of how the drug is eliminated from age 2 months to 18 months. Compared morphine use in infants who received the drug to the group getting placebo. Safety testing for kidney and liver function, breathing measured by continuous oximetry, and any bleeding issues.

DETAILED DESCRIPTION:
Population kinetic analysis of ketorolac stereo-isomer concentrations after single dose given postoperatively in infants aged 2-18 months. Safety assessments of renal and hepatic function tests by blood tests before and after drug administration, urinalysis pre- and post-drug, continuous oximetry before and for 12 hours after drug. Morphine use between active drug groups and placebo group in the first 24 hours after surgery was assessed as a surrogate analgesic measure in these non-verbal infants. A modified infant pain scale was used to assure consistent pain management.

ELIGIBILITY:
Inclusion Criteria:

* Non-prematurely-born infants admitted to hospital following surgery ages 2-18 months, studied by age group 12-18 months, 6-12 months, < 6 months

Exclusion Criteria:

* Bleeding history in infant or family
* Coagulopathy
* Gastrointestinal bleeding history
* Renal or hepatic disease assessed by history and by pre-drug blood tests
* Premature birth (<36 weeks gestation)

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2000-05; Primary Completion 2008-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M. Lynn, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Result] Lynn AM, Bradford H, Kantor ED, Seng KY, Salinger DH, Chen J, Ellenbogen RG, Vicini P, Anderson GD. Postoperative ketorolac tromethamine use in infants aged 6-18 months: the effect on morphine usage, safety assessment, and stereo-specific pharmacokinetics. Anesth Analg. 2007 May;104(5):1040-51, tables of contents. doi: 10.1213/01.ane.0000260320.60867.6c. PMID 17456651
- [Result] Lynn AM, Bradford H, Kantor ED, Andrew M, Vicini P, Anderson GD. Ketorolac tromethamine: stereo-specific pharmacokinetics and single-dose use in postoperative infants aged 2-6 months. Paediatr Anaesth. 2011 Mar;21(3):325-34. doi: 10.1111/j.1460-9592.2010.03484.x. Epub 2010 Dec 29. PMID 21199130

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants less than 18 months of age, having surgery requiring inpatient admission, from 2001 through 2008, with normal renal and liver function, not on chronic medication , not prematurely born, were selected.
Pre-assignment Details: If screening lab studies (blood urea nitrogen [BUN], creatinine, liver transaminase concentrations, urinalysis) were abnormal infants were excluded. If postoperative concerns precluded blood sampling or if sampling intravenous (iv) catheters did not function, infants were excluded.Of 77 infants screened, 51 infants started study
Groups:
- Ketorolac 1 mg/kg Intravenous; Ketorolac 0.5 mg/kg Intravenous; Dextrose 5% in Water (D5W): intravenous infusion over 10 minutes
Period: Overall Study
Arm/Group | Ketorolac 1 mg/kg Intravenous | Ketorolac 0.5 mg/kg Intravenous | Dextrose 5% in Water (D5W)
Started | 22 | 11 | 18
Completed | 22 | 11 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac 1 mg/kg Intravenous | Ketorolac 0.5 mg/kg Intravenous | Dextrose 5% in Water (D5W) | Total
Number analyzed (Participants) | 22 | 11 | 18 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 11 | 18 | 51
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: months] | 8.9 (3.8) | 9.4 (4.2) | 9 (3.8) | 9.1 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants] — while 77 infants were enrolled, exclusions during screening or lack of intravenous access precluding blood sampling eliminated 26 infants. Gender data was not collected for infants not randomized to receive drug or placebo.
  Participants
    Female | 12 | 6 | 8 | 26
    Male | 10 | 5 | 10 | 25
Region of Enrollment [Number; unit: participants]
  United States | 22 | 11 | 18 | 51

OUTCOME MEASURES:

1. Primary Outcome: Clearance of S-ketorolac and R+ Ketorolac in 2-6 Month Old Infants Following Surgery
Description: stereo-isomer specific clearance determined by population-based pharmacokinetic analysis (NONMEM)
Time Frame: 24 hours following surgery
Population: of 25 infants aged 2-6 months enrolled, 11 were excluded. 8 received drug, 6 received placebo; this is a subset of the 77 enrolled infants (aged 2-18 months) of whom 51 completed the study. Infants receiving drug at 0.5 or 1 mg/kg were reported together, since no difference in drug handling was seen.
Measure: Mean (Standard Error); unit: ml/min
Groups:
- S- Ketorolac Clearance: stereo-specific ketorolac isomer concentrations from blood samples collected for 12 hours after ketorolac intravenous administration, analyzed by NONMEM population pharmacokinetic methodology
- R+ Ketorolac Clearance; Placebo: stereo-specific ketorolac isomer concentrations from blood samples collected for 12 hours after ketorolac intravenous administration,analyzed by population pharmacokinetic analysis (NONMEM)
Arm/Group | S- Ketorolac Clearance | R+ Ketorolac Clearance | Placebo
Number analyzed (Participants) | 8 | 8 | 0
ml/min | 30.7 (22.8) | 6.5 (2.2) |

2. Primary Outcome: Central Volume of Distribution for S- and R+ Ketorolac in 2-6 Month Old Infants
Description: stereo-specific ketorolac analysis using population-based analysis (NONMEM)for ketorolac given intravenously 24 hours after surgery in 2-6 month old infants
Time Frame: 24 hours after surgery
Population: infants enrolled but did not complete protocol if abnormal laboratory studies or intravenous catheters were not functioning prior to study drug infusion. Of 77 enrolled, 51 completed study; of the 33 given ketorolac,8 were aged 2-6 months. Doses of 0.5 or 1 mg/kg were handled similarly so reported together.
Measure: Mean (Standard Error); unit: ml
Groups:
- S- Ketorolac Volume Distribution, Central: stereo-specific ketorolac analysis by NONMEM
- R+ Ketorolac Volume Distribution, Central; Placebo: stereo-specific ketorolac analyzed by population kinetic (NONMEM)
Arm/Group | S- Ketorolac Volume Distribution, Central | R+ Ketorolac Volume Distribution, Central | Placebo
Number analyzed (Participants) | 8 | 8 | 0
ml | 1480 (920) | 992 (440) |

3. Primary Outcome: Peripheral Volume of Distribution for S- and R+ Ketorolac in 2-6 Month Old Infants
Description: peripheral volume of distribution for ketorolac stereo-isomers determined by population kinetic analysis (NONMEM)
Time Frame: 24 hours post surgery
Population: 25 infants aged 2-6 months enrolled; 11 excluded for no sampling intravenous access. 8 infants received drug, 6 received placebo. No difference in analysis of doses of 0.5 or 1 mg/kg so reported together.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- S- Ketorolac Volume Distribution, Peripheral: stereo-specific ketorolac analysis by NONMEM
- R+ Ketorolac Volume Distribution, Peripheral; Placebo: stereo-specific ketorolac analyzed by population kinetic (NONMEM)
Arm/Group | S- Ketorolac Volume Distribution, Peripheral | R+ Ketorolac Volume Distribution, Peripheral | Placebo
Number analyzed (Participants) | 8 | 8 | 0
ml | 341 (342) | 658 (207) |

4. Primary Outcome: Half-life of S- and R+ Ketorolac in 2-6 Month Old Infants
Description: half-life calculated from non-compartmental analysis of ketorolac isomers in 2-6 month old infants given intravenous ketorolac following surgery
Time Frame: 24 hours after surgery
Population: total infants enrolled was 77; 26 were excluded before study procedures began. Of 51 infants completing the study, 8 infants aged 2-6 months received drug.No difference in analysis at doses of 0.5 or 1 mg/kg so reported together.
Measure: Mean (Standard Error); unit: min
Groups:
- S- Ketorolac Half-life: stereo-specific ketorolac analysis by NONMEM
- R+ Ketorolac Half-life; Placebo: stereo-specific ketorolac analyzed by population kinetic (NONMEM)
Arm/Group | S- Ketorolac Half-life | R+ Ketorolac Half-life | Placebo
Number analyzed (Participants) | 8 | 8 | 0
min | 67 (33) | 197 (82) |

5. Secondary Outcome: Morphine Use in 2-6 Month Old Infants Given Ketorolac or Placebo Following Surgery
Description: total morphine given intravenously in the 12 hours following receiving intravenous ketorolac or placebo
Time Frame: first day after surgery
Population: 25 infants enrolled but 11 excluded. 8 received ketorolac, 6 placebo. total morphine given over 12 hours following infusion collected
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- Ketorolac 1 or 0.5 mg/kg: infants receiving active drug intravenously after surgery
- Placebo: infants receiving placebo infusion intravenously after surgery
Arm/Group | Ketorolac 1 or 0.5 mg/kg | Placebo
Number analyzed (Participants) | 8 | 6
mg/kg | 0.12 (0.28) | 0.08 (0.12)

6. Secondary Outcome: Percent Time With Room Air Oximetry Saturations Under 90% in 2-6 Month Infants
Description: continuous oximetry monitoring of room air saturation was collected for 12 hours after intravenous infusion of ketorolac or placebo
Time Frame: 12 hours after ketorolac or placebo infusion
Population: 25 infants aged 2-6 months enrolled; 11 excluded. 8 received ketorolac, 6 placebo
Measure: Median (Full Range); unit: percentage of time in 12 h after drug
Groups:
- Ketorolac 1 or 0.5 mg/kg: infants given ketorolac intravenously after surgery
- Placebo: infants given placebo intravenously after surgery
Arm/Group | Ketorolac 1 or 0.5 mg/kg | Placebo
Number analyzed (Participants) | 8 | 6
percentage of time in 12 h after drug | NA [2.1 to 7.3] — Median not calculated due to small sample size | NA [1.9 to 5.1] — Median not calculated due to small sample size

7. Primary Outcome: Clearance of S- and R+ Ketorolac in 6-18 Month Old Infants
Description: stereo-specific ketorolac clearance by population-based analysis (NONMEM)
Time Frame: 24 hours after surgery
Population: 52 infants aged 6-18 months enrolled; 15 excluded for abnormal laboratory results or intravenous sampling catheters that did not allow sampling. 25 infants aged 6-18 months received ketorolac, 12 received placebo. Doses of 0.5 or 1 mg/kg reported together since no difference found in handling.
Measure: Mean (Standard Error); unit: ml/min
Groups:
- S- Ketorolac Clearance: stereo-specific ketorolac analysis by NONMEM
- R+ Ketorolac Clearance; Placebo: stereo-specific ketorolac analyzed by population kinetic (NONMEM)
Arm/Group | S- Ketorolac Clearance | R+ Ketorolac Clearance | Placebo
Number analyzed (Participants) | 25 | 25 | 0
ml/min | 45.3 (12.1) | 7.52 (9.3) |

8. Primary Outcome: Volume of Distribution for Ketorolac Isomers in 6-18 Month Old Infants
Description: population-based kinetic analysis of ketorolac isomers following intravenous infusion in infants after surgery
Time Frame: 24 hours after surgery
Population: of 52 enrolled infants aged 6-18 months, 37 completed the study. Of these, 25 received drug, 12 placebo.Doses of 0.5 or 1 mg/kg showed no difference in handling so reported together.
Measure: Mean (Standard Error); unit: ml
Groups:
- S- Ketorolac Volume Distribution Central: stereo-specific ketorolac analysis by NONMEM
- R+ Ketorolac Volume Distribution Central; Placebo: stereo-specific ketorolac analyzed by population kinetic (NONMEM)
Arm/Group | S- Ketorolac Volume Distribution Central | R+ Ketorolac Volume Distribution Central | Placebo
Number analyzed (Participants) | 25 | 25 | 0
ml | 2320 (14.6) | 1200 (13.6) |

9. Primary Outcome: Ketorolac Stereo-isomer Volume of Distribution Peripheral in 6-18 Month Old Infants
Description: population-based analysis of ketorolac stereo-isomers
Time Frame: 24 hours after surgery
Population: 52 infants aged 6-18 months enrolled; 15 excluded. 25 received ketorolac, 12 received placebo. Drug handling not different at doses of 0.5 or 1 mg/kg so reported together.
Measure: Mean (Standard Error); unit: ml
Arm/Group | S- Ketorolac Volume Distribution, Peripheral | R+ Ketorolac Volume Distribution, Peripheral | Placebo
Number analyzed (Participants) | 25 | 25 | 0
ml | 224 (86) | 828 (13) |

10. Primary Outcome: Half-life of Ketorolac Stereo-isomers in 6-18 Month Old Infants After Surgery
Description: noncompartmental pharmacokinetic analysis of ketorolac stereo-isomers after intravenous infusion in postoperative infants
Time Frame: 24 hours after surgery
Population: 52 infants of the 77 total were aged 6-18 months. 15 were excluded for abnormal laboratory values at screening or for lack of access to draw blood samples. 25 received drug, 12 placebo.Doses 0.5 or 1 mg/kg reported together since no difference in analysis.
Measure: Mean (Standard Deviation); unit: min
Groups:
- S- Ketorolac Half-life: noncompartmental ketorolac analysis
- R+ Ketorolac Half-life; Placebo: noncompartmental analysis of stereo-isomers of ketorolac
Arm/Group | S- Ketorolac Half-life | R+ Ketorolac Half-life | Placebo
Number analyzed (Participants) | 25 | 25 | 0
min | 50.1 (42) | 238 (48) |

11. Secondary Outcome: Total Morphine Use in 6-18 Month Old Infants After Ketorolac or Placebo Intravenous Infusion After Surgery
Description: total amount of morphine given for 12 hours after ketorolac or placebo infusion in 6-18 month old infants after surgery
Time Frame: 24 hours after surgery
Population: 52 infants aged 6-18 months enrolled; 15 excluded. 25 received ketorolac and 12 received placebo infusion after surgery
Measure: Mean (Standard Deviation); unit: mg/kg
Groups:
- Ketorolac 1 or 0.5 mg/kg: infants receiving ketorolac infusion after surgery
- Placebo Infusion: infants receiving placebo infusion after surgery
Arm/Group | Ketorolac 1 or 0.5 mg/kg | Placebo Infusion
Number analyzed (Participants) | 25 | 12
mg/kg | 1.8 (1.5) | 2.2 (1.4)

12. Secondary Outcome: Oximetry Saturation Under 90% After Ketorolac or Placebo Infusion in 6-18 Month Old Infants
Description: continuous oximetry monitoring for 12 hours after ketorolac or placebo intravenous infusion in 6-18 month old infants after surgery
Time Frame: 24 hours after surgery
Population: 52 infants aged 6-18 months enrolled; 15 excluded. 25 received ketorolac, 12 received placebo
Measure: Mean (Standard Deviation); unit: per cent time of 12 hours
Groups:
- Ketorolac 1 or 0.5 mg/kg: infants receiving ketorolac after surgery
Arm/Group | Ketorolac 1 or 0.5 mg/kg | Placebo Infusion
Number analyzed (Participants) | 25 | 12
per cent time of 12 hours | 0.8 (0.8) | 1 (1)

ADVERSE EVENTS:
Time Frame: 24 hours following surgery, monitoring for oximetry, blood loss, renal and liver function tests were done after drug infusion (active drug or placebo)
Arm/Group | Ketorolac 1 mg/kg Intravenous | Ketorolac 0.5 mg/kg Intravenous | Dextrose 5% in Water (D5W)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/11 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No